CLINICAL TRIAL: NCT07133048
Title: Evaluation of Regional Blocks Efficacy in Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, David Harmicar, Principal Investigator, Clinical Hospital Center Rijeka
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHCRijeka
Record Dates: First submitted 2025-06-25; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia
Keywords: anesthesia, conduction;; nerve block;; orthognathic surgery;; pain, postoperative;; postoperative nausea and vomiting;; psychosocial factors
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Levobupivakain 0.25 % (Regional block) (Experimental): Participants receive regional block to II. branch of trigeminal nerve and standard intraoral block to infraorbital nerve.
  Interventions: Procedure: Levobupivakain 0.25 %
- Placebo: NaCl 0.9% (Regional block) (Placebo Comparator): Participants receive regional block to II. branch of trigeminal nerve and standard intraoral block to infraorbital nerve.
  Interventions: Procedure: NaCl 0.9 %

INTERVENTIONS:
Procedure: Levobupivakain 0.25 % — The high tuberosity approach blocks for blockage of II. branch of trigeminal nerve.
  Standard intraoral approach for inferior alveolar nerve block.
  Arms: Experimental: Levobupivakain 0.25 % (Regional block)
Procedure: NaCl 0.9 % — The high tuberosity approach blocks for blockage of II. branch of trigeminal nerve.
  Standard intraoral approach for inferior alveolar nerve block.
  Arms: Placebo: NaCl 0.9% (Regional block)

SUMMARY:
The proposed study, which will be carried out on 72 male and female patients, who have reached bone maturity, are younger than 50 years and underwent orthognathic surgical procedures. Patients will be divided into a study group which will receive a regional block with levobupivacaine and a control group that will receive saline as a placebo. The main hypothesis is that regional analgesia in orthognathic surgery contributes to intraoperative and postoperative analgesia. The aim is to determine the real benefit of regional analgesia in orthognathic surgery and analyze the impact of psychosocial factors on results. Various psychological questionnaires, pain scale and questionnaires for evaluation of postoperative recovery will be used in the research. The results of the research could contribute to a better understanding of regional anesthesia in orthognathic surgery and determine impact of psychosocial factors on pain level and satisfaction with orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* bone deformities for which one of the following surgical procedures is performed: bimaxillary osteotomy, bimaxillary osteotomy with genioplasty, isolated Le Fort I osteotomy, or isolated sagittal osteotomy of the mandible
* patients who have reached skeletal maturity and are under 50 years of age
* patient classified as ASA I and ASA II (American Society of Anesthesiologists).

Exclusion Criteria:

* known allergy to local anesthetics
* refusal to participate in the study
* patients with a cleft of the primary and/or secondary palate
* patients with craniofacial syndromes
* patients who have undergone surgical revision for any reason

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
The amount of analgesics given after surgery | In the first 24 hours after surgery
  The amount of analgesics given after surgery will be measured; patients who have more severe pain will request more analgesics

SECONDARY OUTCOMES:
How mental status (catastrophizing) affects the amount of analgesics taken | The day before surgery participants completed Croatian version of all psychological questionnaires. Analgesics given in the first 24 hours after surgery.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. Number of analgesic in 24 hours.
How mental status (hypervigilance) affects the amount of analgesics taken | The day before surgery participants completed Croatian version of all psychological questionnaires. Analgesics given in the first 24 hours after surgery.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. Number of analgesics in 24 hours.
How mental status (somatosensory amplification) affects the amount of analgesics taken | The day before surgery participants completed Croatian version of all psychological questionnaires. Analgesics given in the first 24 hours after surgery.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. Number of analgesics in 24 hours.
How mental status (anxiety) affects the amount of analgesics taken | The day before surgery participants completed Croatian version of all psychological questionnaires. Analgesics given in the first 24 hours after surgery
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety.Number of analgesics in 24 hours.
Influence of the block on postoperative pain levels | At 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery.
  Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain. The time of the most intense pain level was also examined.
How mental status (catastrophizing) affects the pain level. | The day before surgery participants completed Croatian version of all psychological questionnaires. Pain level at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain.
How mental status (hypervigilance) affects the pain level. | The day before surgery participants completed Croatian version of all psychological questionnaires. Pain level at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain.
How mental status (somatosensory amplification) affects the pain level | The day before surgery participants completed Croatian version of all psychological questionnaires. Pain level at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain.
How mental status (anxiety) affects the pain level | The day before surgery participants completed Croatian version of all psychological questionnaires. Pain level at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery.
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain.
How block affect on postoperative nausea and vomiting | On the first postoperative day, participants completed the PONV questionnaire.
  Participants completed the simplified Postoperative nausea and vomiting (PONV) questionnaire. In this questionnaire with a 0-6 scoring system higher scores indicating more severe symptoms
How mental status (catastrophizing) affects postoperative nausea and vomiting | The day before surgery participants completed Croatian version of all psychological questionnaires. On the first postoperative day, participants completed the PONV questionnaire.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. The simplified Postoperative nausea and vomiting (PONV) questionnaire. In this questionnaire with a 0-6 scoring system higher scores indicating more severe symptoms.
How mental status (hypervigilance) affects postoperative nausea and vomiting | The day before surgery participants completed Croatian version of all psychological questionnaires. On the first postoperative day, participants completed the PONV questionnaire.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. The simplified Postoperative nausea and vomiting (PONV) questionnaire. In this questionnaire with a 0-6 scoring system higher scores indicating more severe symptoms.
How mental status affects (somatosensory amplification) postoperative nausea and vomiting | The day before surgery participants completed Croatian version of all psychological questionnaires. On the first postoperative day, participants completed the PONV questionnaire.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. The simplified Postoperative nausea and vomiting (PONV) questionnaire. In this questionnaire with a 0-6 scoring system higher scores indicating more severe symptoms.
How mental status (anxiety) affects postoperative nausea and vomiting | The day before surgery participants completed Croatian version of all psychological questionnaires. On the first postoperative day, participants completed the PONV questionnaire.
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. The simplified Postoperative nausea and vomiting (PONV) questionnaire. In this questionnaire with a 0-6 scoring system higher scores indicating more severe symptoms.
Influence of the block on the Quality of Life | 2 days after the surgical procedure and at discharge day
  We use the 36-Item Short Form Health Survey (SF-36), as a "Quality of Life" instrument.
  The difference in values between the tested group and the control group was examined. The SF-36 contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
Influence of the level of pain expressed on the VAS scale to the Quality of Life | VAS scale at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery. SF-36 second days after the surgical procedure and at discharge day
  Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain. The SF-36 contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
How mental status (catastrophizing) affects the Quality of Life | The day before surgery participants completed Croatian version of psychological questionnaires. SF-36 second days after the surgical procedure and at discharge day.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. The SF-36 contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
How mental status (hypervigilance) affects the Quality of Life | The day before surgery participants completed Croatian version of psychological questionnaires(BHS). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed SF-36.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. The SF-36 is quality of life marker and contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
How mental status (somatosensory amplification) affects the Quality of Life | The day before surgery participants completed Croatian version of psychological questionnaires(SSAS). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed SF-36.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. The SF-36 is quality of life marker and contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
How mental status (anxiety) affects the Quality of Life | The day before surgery participants completed Croatian version of psychological questionnaires(GAD7). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure)participants completed SF-36.
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. The SF-36 is quality of life marker and contains 36 items and measures perceived health status by assessing eight health components each scoring from 0 to 100, with higher scores indicating better health status.
Influence of the block on the Quality of Recovery | The first day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed Croatian version of QoR-40 questionnaire.
  The QoR-40 is marker of postoperative recovery and score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
Influence of the block on the satisfaction with the surgical procedure | Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction
Influence of the level of pain expressed on the VAS scale to the Quality of Recovery (QoR-40) | VAS scale at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery. Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed QoR-40.
  Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain. The QoR-40 score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
How mental status (catastrophizing) affects the Quality of Recovery | The day before surgery participants completed Croatian version of psychological questionnaire (PCS). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed QoR-40.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. The QoR-40 score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
How mental status (hypervigilance) affects the Quality of Recovery | The day before surgery participants completed Croatian version of all psychological questionnaires (BHS). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed QoR-40.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. The QoR-40 score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
How mental status (somatosensory amplification) affects the Quality of Recovery | The day before surgery participants completed Croatian version of psychological questionnaires (SSAS). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed QoR-40.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. The QoR-40 score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
How mental status (anxiety) affects the Quality of Recovery | The day before surgery participants completed Croatian version of psychological questionnaires (GAD7). Second day after the surgical procedure and at discharge day (an average of third day after surgical procedure) participants completed QoR-40.
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. The QoR-40 score ranges from 40 (indicating a poor quality of recovery) to 200 (indicating an excellent quality of recovery).
Influence of the level of pain expressed on the VAS scale to the satisfaction with the surgical procedure | VAS scale at 1 hour, 3 hours, 5 hours, 7 hours, 9 hours, 12 hours, and 24 hours after the end of the surgery. Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  Postoperative pain levels were assessed using the VAS scale (0-10). Higher scores indicating greater pain. For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction.
How mental status (catastrophizing) affects the satisfaction with the surgical procedure | The day before surgery participants completed Croatian version of psychological questionnaires. Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  Pain Catastrophizing Scale (PCS), total score ranges from 0 to 52, with higher scores indicating more severe pain catastrophizing. For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction
How mental status (hypervigilance) affects the satisfaction with the surgical procedure | The day before surgery participants completed Croatian version of psychological questionnaires. Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  Brief Hypervigilance Scale (BHS), range from 0 to 20, with higher scores indicating greater hypervigilance. For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction
How mental status (somatosensory amplification) affects the satisfaction with the surgical procedure | The day before surgery participants completed Croatian version of psychological questionnaires. Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  Somatosensory Amplification Scale (SSAS), ranges from 10 to 50, with higher scores indicating greater somatosensory amplification. For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction
How mental status (anxiety) affects the satisfaction with the surgical procedure | The day before surgery participants completed Croatian version of psychological questionnaires. Two months after the surgical procedure, the patient completed the SSQ-8 questionnaire.
  General Anxiety Disorder-7 (GAD7) scale has a total score range of 0 to 21 and scores are categorized as follows: 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. For a general assessment of satisfaction with the surgical procedure, the Surgical Satisfaction Questionnaire (SSQ-8) was used.SSQ-8 ranges from 0 to 100, where 100 represents the highest level of satisfaction

OTHER OUTCOMES:
The length of hospital stay after the surgical procedure | The day count starts from the first postoperative day until the day of discharge from the hospital day (an average of third day after surgical procedure).
  Number of days spent in hospital after the procedure
Complications and side effects | Recording of complications begins from the time the regional block is administered until the day of discharge from the hospital day (an average of third day after surgical procedure).
  All complication of surgery and preemptive block

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Maxillofacial surgery, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All data included in the research can be shared. Except for the personal data of the participants.
Supporting Information: ICF